CLINICAL TRIAL: NCT02388217
Title: The Effect of Cannabis on Pain and Related Quality Of Life Outcomes In Chronic Pain: A Prospective Open-Label Study
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Elyad Davidson, MD, Hadassah Medical Organization
Other Study IDs: 07419-10-HMO
Record Dates: First submitted 2014-04-06; First posted 2015-03-13 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pain
Keywords: chronic pain; cannabis; Approved for cannabis treatment by Israeli ministry of health; Unrelieved chronic pain
MeSH Terms: conditions — Chronic Pain; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the current study is to prospectively assess the effect of cannabis on pain and functional outcomes in a large group of patients with chronic pain.

DETAILED DESCRIPTION:
This is a prospective, observational, open-label study carried out at the ambulatory pain clinic of Hadassah-Hebrew University Medical Center Pain Relief Unit.

Study population: Patients suffering from chronic pain that has not been relieved with other analgesic medications, who are eligible for treatment with medical cannabis (cigarettes, oil or cookies) following approval of Israeli Ministry of health.The patients will receive a prescription to be dispensed at pre-approved cannabis distribution points by a certified provider.

In this study, the efficacy of the cannabis treatment on pain and related quality of life (QoL) outcomes will be assessed by administering the S-TOPS questionnaire (Haroutiunian, Pain 2012), and the Brief Pain Inventory (BPI) before the treatment (baseline), and on expected follow-up visits at approximately 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Chronic pain, with duration of 3 months or longer
* Lack of satisfactory analgesic response or intolerable adverse effects with at least two analgesics from 2 different drug classes at full dose.

Exclusion Criteria:

* Inability to read and understand the informed consent form.
* History of drug abuse/dependence
* Psychiatric co morbidity (or history) of schizophrenia or acute psychosis.
* Family history of schizophrenia.
* Psychologist evaluation of high abuse risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patients with lack of satisfactory analgesic response or intolerable adverse effects with at least two analgesics from 2 different drug classes at full dose. Eligible for cannabis treatment following Israeli Ministry of Health approval.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-03-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the S-TOPS pain symptom scale | 1 year
  The primary outcome is pain reduction (change from baseline) assessed by the Pain Symptom scale of the S-TOPS instrument

SECONDARY OUTCOMES:
Change from baseline on S-TOPS physical disability scales | 6 and 12 months
Change from baseline on S-TOPS emotional/social disability scales | 6 and 12 months
Change from baseline on S-TOPS satisfaction scales | 6 and 12 months
Change from baseline on SLP9 sleep disability scale | 6 and 12 months
Change from baseline on BPI severity/interference scales | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel